CLINICAL TRIAL: NCT05652179
Title: Pretreatment with Stellate Ganglion Block Reduces the Incidence and Severity of Cardiac Surgery-Associated Acute Kidney Injury
Brief Title: SGB Reduces the Incidence and Severity of CSA-AKI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yangzhou University (Other)
Responsible Party: Principal Investigator, Zhuan Zhang, Principal Investigator, Yangzhou University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 20221107
Record Dates: First submitted 2022-11-06; First posted 2022-12-15 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2024-03

CONDITIONS: Stellate Ganglion Block
Keywords: Stellate ganglion block; Cardiac surgery; Acute kidney injury; Sympathetic nerve; Renal artery; Resistance index
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Stellate ganglion block (Experimental): For patients in Group S, left SGB was performed after the first TEE examination. The patient's head was tilted to the right. A high-frequency probe (6-13 MHz) was placed between the C6 and C7 transverse processes to obtain the best image of the longus colli muscle. After iodine disinfection, a 22-G atraumatic needle for peripheral nerve blocks (B. Braun Melsungen AG, Melsungen, Germany) was used to puncture the site posterior to the left carotid artery and on the surface of the longus colli muscle via an in-plane technique. Then,5 mL of 0.375% ropivacaine hydrochloride injection was administered provided that no blood, cerebrospinal fluid, or gas was suctioned out
  Interventions: Drug: Stellate ganglion block
- Control (No Intervention): Patients in Group C did not undergo the SGB procedure.

INTERVENTIONS:
Drug: Stellate ganglion block — After the induction of general anesthesia and before the start of the surgery,ultrasound-guided stellate ganglion block is performed, injecting 5 ml of 0.375% ropivacaine.
  Arms: Stellate ganglion block

SUMMARY:
The incidence of acute kidney injury after cardiopulmonary bypass cardiac surgery is high, which increases postoperative mortality and is not conducive to the prognosis of patients. Stellate ganglion blocks increase renal blood flow, reduce inflammation and stress, and protect the heart muscle. In this study, stellate ganglion block was used to promote rapid recovery of kidney function after cardiopulmonary bypass cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Patients of any gender were eligible provided they were between the ages of 18 and 80 years;
2. American Society of Anesthesiologists (ASA) class of Ⅲ or IV.

Exclusion Criteria:

1. emergency cardiac surgery；
2. major vascular surgery；
3. non-sinus rhythm, reoperation；
4. contraindications for TEE or SGB；
5. abnormal preoperative renal function；
6. severe preoperative heart failure with left ventricular ejection fraction < 30%, multi-organ dysfunction；
7. and severe infection requiring continuous antibiotic treatment;
8. enrolled in another clinical trial.

Elimination criteria:

1. incomplete follow-up data;
2. withdrawal during the procedure;
3. SGB failure or complications;
4. insufficient ultrasonographic imaging of the left renal artery on TEE;
5. repeated CPB during surgery;
6. need for cardiac assist devices (extracorporeal membrane oxygenation, intra-aortic balloon pump, or ventricular assist devices) after CPB completion.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 396 (Actual)
Dates: Start 2023-01-10 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
The incidence and severity of CSA-AKI | From the end of surgey to postoperative day 7
  Postoperative serum creatinine was detected once a day from the patient's arrival in the ICU until postoperative day 7. The severity of CSA-AKI was graded by the change in the plasma creatinine levels, according to the Kidney Disease: Improving Global Outcomes (KDIGO) criteria

SECONDARY OUTCOMES:
Changes of intraoperative left RBF parameters | 5 minutes after general anesthesia induction,15 minutes after the SGB procedure in Group S and 20 minutes after the completion of the first TEE examination in Group C, and 30 minutes after the end of CPB
  The peak systolic velocity (PSV), end-diastolic velocity (EDV), mean blood flow velocity (V-mean), the diameter of the left renal artery (RAD)and velocity time integral (VTI) of the left renal artery were measured
Changes of perioperative BNP, CK-MB, IL-6, CRP, IL-18, and norepinephrine levels | preoperatively, Immediately after the surgery,the first day after surgery,the second day after surgery, and the seventh day after surgery
  Venous blood samples were collected to test BNP (Brain natriuretic peptide), CK-MB (Creatine kinase isoenzymes), kidney injury molecule-1 (KIM-1), interleukin (IL)-6, C-reactive protein (CRP), IL-18, and norepinephrine levels.
Comparison of recovery indicators between the 2 groups | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  The duration of mechanical ventilation in the ICU, length of ICU stay, length of postoperative hospitalization in the ward, and in-hospital mortality were recorded
Hemodynamic changes during surgery. | after radial artery cannulation,5 min after general anesthesia induction,15 min after the SGB procedure ,30 min after CPB initiation,30 min after the end of CPB,and the end of surgery.
  The MAP from the radial artery,HR,CVP, and cardiac output.

CONTACTS AND LOCATIONS:
Locations (1):
- the Affiliated Hospital of Yangzhou University, Yangzhou University, Yangzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No